CLINICAL TRIAL: NCT03174444
Title: Small Media Interventions to Increase Colorectal Cancer Screening Among Chinese Americans
Acronym: SMILES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); NICOS Chinese Health Coalition (Unknown); Chinese Community Health Resource Center (Other); Northeast Medical Services (Unknown); Chinese Hospital Clinics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 174519; 3U48DP004998-03S6 (NIH)
Record Dates: First submitted 2017-05-30; First posted 2017-06-02 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Colorectal Cancer; Cancer Screening
Keywords: Chinese American; Asian American; Colorectal cancer screening; Print materials
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Individual randomized controlled trial with two arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Small Media (Experimental): Participants receive bilingual brochures and access to bilingual website about colorectal cancer screening.
  Interventions: Behavioral: Small Media
- Control (No Intervention): Participants receive no information about colorectal cancer screening from the study during the intervention period, but may receive usual care from health care provider.

INTERVENTIONS:
Behavioral: Small Media — Bilingual brochures and access to bilingual website
  Arms: Small Media

SUMMARY:
There have been few studies of small media interventions to promote colorectal cancer screening among Chinese Americans. Based on the results of strong preliminary studies on the promotion of colorectal cancer screening among Asian American populations, this community-academic research team propose to develop a culturally and linguistically appropriate traditional small media print brochure and a novel small media electronic audio-visual application accessible through mobile applications and through a website to promote CRC screening in English, Cantonese, and Mandarin. The team will test in a randomized controlled trial in 3 healthcare systems the efficacy of a combination of these small media interventions and a mailed patient reminder compared to usual care on increasing CRC screening among Chinese American patients.

DETAILED DESCRIPTION:
Chinese Americans are the largest group of Asian Americans, the fastest growing racial population in the U.S. Colorectal cancer is the second most common cancer among Chinese Americans. Screening reduces colorectal cancer mortality and is cost-effective but remains underutilized. Asian Americans and Chinese Americans are less likely than non-Hispanic whites to be screened for colorectal cancer. Factors associated with lack of screening among Asian Americans include recent immigration, lower education, lower English fluency, lack of knowledge, patient-physician language discordance, and lack of physician recommendation.

Although small media and client-reminders are effective in increasing colorectal cancer screening in the general population, no randomized controlled trial has assessed the effect of such interventions on Chinese Americans, particularly those who are limited English proficient. Building on an established community-based participatory research network and strong preliminary studies, the team propose to develop a culturally and linguistically appropriate booklet (small print media) and an audio-visual application accessible through mobile devices and a website (small electronic media) to promote screening. Through an innovative approach that links community organizations that have cultural and linguistic expertise to healthcare systems that have many Chinese American patients, the investigators will test the effect of combining these small media materials and a mailed patient reminder on the rate of screening for colorectal cancer screening among Chinese Americans in this Small Media Interventions for Limited English Speakers (SMILES). The investigators have developed English and Chinese (Cantonese and Mandarin) small print and electronic media materials to promote colorectal cancer screening among Chinese Americans. This RCT will compare the efficacy of a combination of mailed patient reminder and small print and electronic media versus usual care among Chinese American patients who are not up-to-date for colorectal cancer screening recruited from 3 healthcare systems in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Not up-to-date for colorectal cancer screening; self-identified as Chinese or Chinese American, or Asian who speak Chinese, or Asian born in China.

Exclusion Criteria:

* Not eligible for colorectal cancer screening for any reason.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1707 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Colorectal Cancer Screening | 9 months
  Up-to-date receipt of any colorectal cancer screening

CONTACTS AND LOCATIONS:
Overall Officials: Tung Nguyen, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No